CLINICAL TRIAL: NCT02498652
Title: A Phase 2a, Randomized, Open-Label Study to Evaluate the Pharmacodynamic Effects and Safety of RDEA3170 Administered in Combination With Allopurinol Compared With Allopurinol Administered Alone in Adult Subjects With Gout
Brief Title: Phase 2a RDEA3170 and Allopurinol Combination Study in Gout Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDEA3170-206
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — verinurad; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RDEA3170 2.5 mg, 7.5 mg and 15 mg (Experimental): RDEA3170 2.5 mg, 7.5 mg and 15 mg once daily (qd) in combination with allopurinol 300 mg (qd and twice daily (bid))
  Interventions: Drug: RDEA3170 2.5 mg; Drug: allopurinol 300 mg
- RDEA3170 5 mg, 10 mg and 20 mg (Experimental): RDEA3170 5 mg, 10 mg 20 mg qd in combination with allopurinol 300 mg (qd and bid)
  Interventions: Drug: RDEA3170 2.5 mg; Drug: allopurinol 300 mg

INTERVENTIONS:
Drug: RDEA3170 2.5 mg — Cohort 1: RDEA3170 2.5 mg, 7.5 mg (2.5 mg × 3 tablets), and 15 mg (2.5 mg × 6 tablets).
  Cohort 2: RDEA3170 5 mg (2.5 mg × 2 tablets), 10 mg (2.5 mg × 4 tablets), and 20 mg (2.5 mg × 8 tablets).
Drug: allopurinol 300 mg — allopurinol 300 mg, allopurinol 600 mg (300 mg x 2 tablets)

SUMMARY:
This is a Phase 2a, randomized, open-label, multicenter study to assess the pharmacodynamic (PD) effects of RDEA3170 administered in combination with allopurinol compared with allopurinol administered alone in adult subjects with gout.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures and the risks involved and is willing to provide written informed consent before the first study-related activity.
* Subject meets one or more criteria for the diagnosis of gout as per the American Rheumatism Association Criteria for the Classification of Acute Arthritis of Primary Gout.
* Subject has a body weight ≥ 50 kg (110 lbs.) and a body mass index ≥ 18 and ≤ 45 kg/m2.
* Subject has a Screening serum urate level ≥ 8 mg/dL.
* Subject is free of any clinically significant disease or medical condition, per the Investigator's judgment.

Exclusion Criteria:

* Subject is unable to take colchicine for gout flare prophylaxis.
* Subject has a history or suspicion of kidney stones.
* Subject has any gastrointestinal disorder that affects motility and/or absorption.
* Subject had unstable angina, New York Heart Association class III or IV heart failure, ischemic heart disease, stroke, or deep venous thrombosis within 12 months prior to Day 1; or subject is currently receiving anticoagulants.
* Subject has Screening laboratory parameters that are outside the normal limits and are considered clinically significant by the Investigator.
* Subject has an estimated creatinine clearance < 60 mL/min calculated by the Cockcroft-Gault formula using ideal body weight during the Screening period.
* Subject is taking losartan, fenofibrate, guaifenesin, or sodium-glucose linked transporter-2 inhibitors; chronic and stable doses are permitted if doses are stable for at least 14 days prior to study medication dosing.
* Subject is unable or unwilling to comply with the study requirements or has a situation or condition that, in the opinion of the Investigator, may interfere with participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2015-11-19 (Actual); Study Completion 2016-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Hall, MD, Study Director — Ardea Biosciences, Inc.
Locations (4):
- United States (4):
  - Anaheim, California
  - DeLand, Florida
  - South Miami, Florida
  - Dallas, Texas

REFERENCES:
- [Derived] Fleischmann R, Winkle P, Miner JN, Yan X, Hicks L, Valdez S, Hall J, Liu S, Shen Z, Gillen M, Hernandez-Illas M. Pharmacodynamic and pharmacokinetic effects and safety of verinurad in combination with allopurinol in adults with gout: a phase IIa, open-label study. RMD Open. 2018 Feb 8;4(1):e000584. doi: 10.1136/rmdopen-2017-000584. eCollection 2018. PMID 29531784

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 subjects were randomized.
Pre-assignment Details: Forty-one subjects were randomized and received at least 1 dose of randomized study medication; 20 subjects in Cohort 1 and 21 subjects in Cohort 2. Subjects were randomized into 1 of 8 sequences across the 2 cohorts (20 subjects each) in a 1:1 ratio.A total of 40 subjects completed the study.
Groups:
- Cohort 1: Allopurinol 300 mg once daily (qd), 600 mg qd, RDEA3170 2.5 mg qd, 15 mg qd and 7.5 mg qd
- Cohort 2: Allopurinol 300 mg qd, 600 mg (300 mg bid), RDEA3170 5 mg qd, 20 mg qd and 10 mg qd
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 20 | 21
Completed | 20 | 20 (One subject was withdrawn due to noncompliance/protocol violation)
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50 (12.7) | 48 (10.9) | 49 (11.7)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 1 | 0 | 1
  Female | 19 | 21 | 40
Region of Enrollment [Number; unit: Participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1 - Maximum Percentage (%) Change in Serum Urate of Multiple-dose RDEA3170 Administered in Combination With Allopurinol (Emax, CB (%))
Description: Pharmacodynamics (PD) profile of multiple-dose RDEA3170 administered in combination with allopurinol (Cohort 1)
Time Frame: Screening, Days -1 , 1, 7, 14, 21, 28, and 35 (Pre-dose and Post-dose)
Measure: Mean (Standard Error); unit: Maximum Percentage (%) Change
Groups:
- Treatment A1: Allopurinol 300 mg qd
- Treatment A2q: Allopurinol 600 mg qd
- Treatment A2b: Allopurinol 600 mg (300 mg bid)
- Treatment R1: Allopurinol 300 mg qd + RDEA3170 2.5 mg qd
- Treatment R3: Allopurinol 300 mg qd + RDEA3170 7.5 mg qd
- Treatment R5: Allopurinol 300 mg qd + RDEA3170 15 mg qd
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R1 | Treatment R3 | Treatment R5
Number analyzed (Participants) | 20 | 10 | 10 | 20 | 20 | 20
Maximum Percentage (%) Change | -40.2 (3.29) | -55.0 (4.96) | -56.8 (4.52) | -48.1 (2.91) | -61.0 (2.59) | -69.5 (2.09)

2. Primary Outcome: Cohort 1 - Concentration of Serum Urate at 24hr of Multiple-dose RDEA3170 Administered in Combination With Allopurinol.
Description: Pharmacodynamics (PD) profile of multiple-dose RDEA3170 administered in combination with allopurinol (Cohort 1)
Time Frame: Screening, Days -1 , 1, 7, 14, 21, 28, and 35 (Pre-dose and Post-dose)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R1 | Treatment R3 | Treatment R5
Number analyzed (Participants) | 20 | 10 | 10 | 20 | 20 | 20
mg/dL | 5.8 (0.24) | 4.8 (0.38) | 4.0 (0.39) | 5.5 (0.24) | 4.6 (0.22) | 3.8 (0.18)

3. Primary Outcome: Cohort 1 - Renal Xanthine Excretion at 0-24hr of Multiple-dose RDEA3170 Administered in Combination With Allopurinol (AeXO, CB (%))
Description: Pharmacodynamics (PD) profile of multiple-dose RDEA3170 administered in combination with allopurinol (Cohort 1)
Time Frame: Screening, Days -1 , 1, 7, 14, 21, 28, and 35 (Pre-dose and Post-dose)
Measure: Mean (Standard Error); unit: Percentage (%) Change
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R1 | Treatment R3 | Treatment R5
Number analyzed (Participants) | 20 | 10 | 10 | 20 | 20 | 20
Percentage (%) Change | 1065 (138) | 1827 (252) | 2633 (255) | 899 (116) | 958 (128) | 827 (106)

4. Primary Outcome: Cohort 1 - Renal Hypoxanthine Excretion at 0-24hr of Multiple-dose RDEA3170 Administered in Combination With Allopurinol (AeHXO, CB (%))
Description: Pharmacodynamics (PD) profile of multiple-dose RDEA3170 administered in combination with allopurinol (Cohort 1)
Time Frame: Screening, Days -1 , 1, 7, 14, 21, 28, and 35 (Pre-dose and Post-dose)
Measure: Mean (Standard Error); unit: Percentage (%) Change
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R1 | Treatment R3 | Treatment R5
Number analyzed (Participants) | 20 | 10 | 10 | 20 | 20 | 20
Percentage (%) Change | 400 (74.6) | 517 (106) | 827 (136) | 310 (55.5) | 311 (51.8) | 305 (54.7)

5. Primary Outcome: Cohort 2 - Maximum Percentage (%) Change in Serum Urate of Multiple-dose RDEA3170 Administered in Combination With Allopurinol (Emax, CB (%))
Description: Pharmacodynamics (PD) profile of multiple-dose RDEA3170 administered in combination with allopurinol (Cohort 2)
Time Frame: Screening, Days -1 , 1, 7, 14, 21, 28, and 35 (Pre-dose and Post-dose)
Measure: Mean (Standard Error); unit: Maximum Percentage (%) Change
Groups:
- Treatment R2: Allopurinol 300 mg qd + RDEA3170 5 mg qd
- Treatment R4: Allopurinol 300 mg qd + RDEA3170 10 mg qd
- Treatment R6: Allopurinol 300 mg qd + RDEA3170 20 mg qd
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R2 | Treatment R4 | Treatment R6
Number analyzed (Participants) | 20 | 10 | 10 | 20 | 20 | 20
Maximum Percentage (%) Change | -39.3 (1.78) | -54.4 (4.50) | -50.3 (4.15) | -57.8 (1.61) | -66.0 (1.86) | -73.2 (1.75)

6. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: Cmax of Allopurinol alone or in combination with RDEA3170
Time Frame: Day 7, 14, 21, 28 and 35 (predose through 24 hours postdose)
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Treatment A1: Allopurinol 300 mg qd (Cohorts 1 and 2)
- Treatment A2q: Allopurinol 600 mg (qd) (Cohorts 1 and 2)
- Treatment A2b: Allopurinol 600 mg (300 mg bid) (Cohorts 1 and 2)
- Treatment R1: Allopurinol 300 mg qd + RDEA3170 2.5 mg qd (Cohort 1)
- Treatment R2: Allopurinol 300 mg qd + RDEA3170 5 mg qd (Cohort 2)
- Treatment R3: Allopurinol 300 mg qd + RDEA3170 7.5 mg qd (Cohort 1)
- Treatment R4: Allopurinol 300 mg qd + RDEA3170 10 mg qd (Cohort 2)
- Treatment R5: Allopurinol 300 mg qd + RDEA3170 15 mg qd (Cohort 1)
- Treatment R6: Allopurinol 300 mg qd + RDEA3170 20 mg qd (Cohort 2)
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R1 | Treatment R2 | Treatment R3 | Treatment R4 | Treatment R5 | Treatment R6
Number analyzed (Participants) | 40 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
µg/mL | 1.18 [1.03 to 1.36] | 2.43 [1.94 to 3.04] | 1.19 [0.997 to 1.42] | 1.16 [0.911 to 1.47] | 1.16 [0.937 to 1.43] | 1.14 [0.905 to 1.44] | 1.11 [0.928 to 1.33] | 1.12 [0.877 to 1.44] | 1.26 [1.02 to 1.56]
Statistical Analysis 1: Comparison: Treatment A1 vs Treatment R1; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects; Geometric Least Squares Mean Ratio (%) = 103, 90% CI 2-sided [90.7 to 117]
Statistical Analysis 2: Comparison: Treatment A1 vs Treatment R2; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects; Geometric Least Squares Mean Ratio (%) = 92.6, 90% CI 2-sided [78.1 to 110]
Statistical Analysis 3: Comparison: Treatment A1 vs Treatment R3; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 102, 90% CI 2-sided [85.7 to 120]
Statistical Analysis 4: Comparison: Treatment A1 vs Treatment R4; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 88.9, 90% CI 2-sided [78.4 to 101]
Statistical Analysis 5: Comparison: Treatment A1 vs Treatment R5; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 100, 90% CI 2-sided [87.7 to 114]
Statistical Analysis 6: Comparison: Treatment A1 vs Treatment R6; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 101, 90% CI 2-sided [85.5 to 119]

7. Secondary Outcome: Time of Occurrence of Maximum Observed Concentration (Tmax)
Description: Tmax of Allopurinol alone or in combination with RDEA3170
Time Frame: Day 7, 14, 21, 28 and 35 (predose through 24 hours postdose)
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R1 | Treatment R2 | Treatment R3 | Treatment R4 | Treatment R5 | Treatment R6
Number analyzed (Participants) | 40 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
hr | 1.50 [0.500 to 6.02] | 2.98 [0.983 to 4.00] | 2.02 [0.500 to 8.00] | 2.01 [0.967 to 6.00] | 2.49 [0.500 to 3.97] | 1.73 [0.500 to 6.00] | 2.98 [0.500 to 6.02] | 1.73 [0.500 to 6.00] | 1.97 [0.500 to 4.03]

8. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero up to 24 Hours Postdose (AUC 0-24)
Description: AUC 0-24 of Allopurinol alone or in combination with RDEA3170
Time Frame: Day 7, 14, 21, 28 and 35 (predose through 24 hours postdose)
Measure: Geometric Mean (95% Confidence Interval); unit: µg·hr/mL
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R1 | Treatment R2 | Treatment R3 | Treatment R4 | Treatment R5 | Treatment R6
Number analyzed (Participants) | 40 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
µg·hr/mL | 3.94 [3.52 to 4.42] | 11.0 [8.87 to 13.7] | 8.64 [7.13 to 10.5] | 4.06 [3.24 to 5.10] | 4.10 [3.53 to 4.77] | 3.81 [3.13 to 4.64] | 3.83 [3.15 to 4.65] | 3.88 [3.15 to 4.77] | 3.82 [3.27 to 4.46]

9. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Sampling Timepoint (AUC Last)
Description: AUC last of Allopurinol alone or in combination with RDEA3170
Time Frame: Day 7, 14, 21, 28 and 35 (predose through 24 hours postdose)
Measure: Geometric Mean (95% Confidence Interval); unit: µg·hr/mL
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R1 | Treatment R2 | Treatment R3 | Treatment R4 | Treatment R5 | Treatment R6
Number analyzed (Participants) | 40 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
µg·hr/mL | 3.70 [3.28 to 4.18] | 10.9 [8.74 to 13.5] | 4.25 [3.57 to 5.07] | 3.59 [2.87 to 4.49] | 3.76 [3.20 to 4.41] | 3.71 [3.04 to 4.54] | 3.53 [2.84 to 4.39] | 3.74 [3.21 to 4.34] | 3.74 [3.21 to 4.34]
Statistical Analysis 1: Comparison: Treatment A1 vs Treatment R1; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 100, 90% CI 2-sided [94.3 to 107]
Statistical Analysis 2: Comparison: Treatment A1 vs Treatment R2; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 98.0, 90% CI 2-sided [90.4 to 106]
Statistical Analysis 3: Comparison: Treatment A1 vs Treatment R3; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 104, 90% CI 2-sided [94.5 to 114]
Statistical Analysis 4: Comparison: Treatment A1 vs Treatment R4; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 92.0, 90% CI 2-sided [86.7 to 97.7]
Statistical Analysis 5: Comparison: Treatment A1 vs Treatment R5; Test type: Non-Inferiority — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 98.9, 90% CI 2-sided [91.0 to 107]
Statistical Analysis 6: Comparison: Treatment A1 vs Treatment R6; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Mixed Models Analysis; Fixed effect for treatment and random effects for subjects. GLMSRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 97.5, 90% CI 2-sided [92.8 to 102]

10. Secondary Outcome: Apparent Terminal Half-life (t1/2)
Description: t1/2 of Allopurinol alone or in combination with RDEA3170
Time Frame: Day 7, 14, 21, 28 and 35 (predose through 24 hours postdose)
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R1 | Treatment R2 | Treatment R3 | Treatment R4 | Treatment R5 | Treatment R6
Number analyzed (Participants) | 40 | 20 | 20 | 20 | 20 | 20 | 20 | 20 | 20
hr | 1.21 [1.14 to 1.27] | 1.47 [1.33 to 1.62] | 1.25 [1.13 to 1.38] | 1.20 [1.10 to 1.30] | 1.14 [1.03 to 1.25] | 1.17 [1.10 to 1.25] | 1.16 [1.08 to 1.24] | 1.13 [1.04 to 1.22] | 1.13 [1.03 to 1.24]

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Time Frame: 11 weeks
Measure: Number; unit: Number of participants
Groups:
- Cohort 1: RDEA3170 2.5 mg, 7.5 mg and 15 mg qd in combination with allopurinol 300 mg (qd and bid)
- Cohort 2: RDEA3170 5 mg, 10 mg 20 mg qd in combination with allopurinol 300 mg (qd and bid)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 20 | 21
Number of participants | 6 | 6

12. Primary Outcome: Cohort 2 - Concentration of Serum Urate at 24hr of Multiple-dose RDEA3170 Administered in Combination With Allopurinol.
Description: Pharmacodynamics (PD) profile of multiple-dose RDEA3170 administered in combination with allopurinol (Cohort 2)
Time Frame: Screening, Days -1 , 1, 7, 14, 21, 28, and 35 (Pre-dose and Post-dose)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R2 | Treatment R4 | Treatment R6
Number analyzed (Participants) | 20 | 10 | 10 | 20 | 20 | 20
mg/dL | 6.2 (0.22) | 5.0 (0.61) | 4.6 (0.33) | 4.8 (0.22) | 4.1 (0.22) | 3.5 (0.20)

13. Primary Outcome: Cohort 2 - Renal Xanthine Excretion at 0-24hr of Multiple-dose RDEA3170 Administered in Combination With Allopurinol (AeXO, CB (%))
Description: Pharmacodynamics (PD) profile of multiple-dose RDEA3170 administered in combination with allopurinol (Cohort 2)
Time Frame: Screening, Days -1 , 1, 7, 14, 21, 28, and 35 (Pre-dose and Post-dose)
Measure: Mean (Standard Error); unit: Percentage (%) Change
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R2 | Treatment R4 | Treatment R6
Number analyzed (Participants) | 20 | 10 | 10 | 20 | 20 | 20
Percentage (%) Change | 952 (77.2) | 2027 (203) | 2138 (164) | 812 (76.3) | 797 (65.7) | 816 (71.1)

14. Primary Outcome: Cohort 2 - Renal Hypoxanthine Excretion at 0-24hr of Multiple-dose RDEA3170 Administered in Combination With Allopurinol (AeHXO, CB (%))
Description: Pharmacodynamics (PD) profile of multiple-dose RDEA3170 administered in combination with allopurinol (Cohort 2)
Time Frame: Screening, Days -1 , 1, 7, 14, 21, 28, and 35 (Pre-dose and Post-dose)
Measure: Mean (Standard Error); unit: Percentage (%) Change
Arm/Group | Treatment A1 | Treatment A2q | Treatment A2b | Treatment R2 | Treatment R4 | Treatment R6
Number analyzed (Participants) | 20 | 10 | 10 | 20 | 20 | 20
Percentage (%) Change | 372 (33.9) | 645 (76.9) | 681 (63.9) | 268 (24.1) | 267 (23.4) | 286 (25.6)

ADVERSE EVENTS:
Time Frame: 11 Weeks.
Description: Total # Affected by any Other Adverse Event includes subjects who may appear more than once; Other Adverse Events were reported for 6 subjects in Cohort 1 and 6 subjects in Cohort 2.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/21
Other Adverse Events (participants affected / at risk) | 6/20 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=20) | Cohort 2 (N=21)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=20) | Cohort 2 (N=21)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Reliable urine uric acid values were not obtained due to sample processing errors, and this has resulted in the inability to assess the PD effects of RDEA3170 and/or allopurinol in urine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.